CLINICAL TRIAL: NCT03497936
Title: Marketability of a Technology-based Intervention to Increase HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Prevention, LLC (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DP006291 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-04-13 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Human Papilloma Virus
Keywords: vaccine narratives; HPV prevention; vaccine promotion

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of two arms (intervention, no intervention). Intervention participants receive Women's Stories. No intervention participants receive treatment as usual. All participants are administered a pretest and two post tests, and clinical records are examined for vaccination outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women's Stories (Experimental): Participants in this group will be randomly assigned to use the Women's Stories intervention.
  Interventions: Behavioral: Women's Stories
- Programming as usual (No Intervention): Participants in this group will be randomly assigned participate in their usual programming.

INTERVENTIONS:
Behavioral: Women's Stories — Women's Stories is a brief, HPV vaccination promotion intervention. It presents vaccine information and videos of HPV vaccine decision making. It also includes follow up vaccine reminder text messages.
  Arms: Women's Stories

SUMMARY:
The overall goal of this SBIR Phase II project is to reduce cancer rates by marketing a brief, easily implemented technology-based intervention that increases human papillomavirus (HPV) vaccination among Planned Parenthood and other clients. The intervention's innovative technology allows for the investigators' narrative videos to be presented along will reminder texts. It will be evaluated for use in waiting rooms and promises to overcome vaccination barriers among high risk but underserved low SES and minority populations.

DETAILED DESCRIPTION:
The purpose of this Phase II research project is to evaluate and market an innovative health message intervention to increase uptake of the human papillomavirus (HPV) vaccine and reduce women's cervical cancer risk through partnership with Planned Parenthood. The overall aim is to reach a broad population through Planned Parenthood, the nation's leading sexual and reproductive health care center, especially among low socioeconomic status (SES) and historically underserved populations. Despite an overall increase in vaccination and reduction in HPV-related infections in younger populations targeted by previous health promotion efforts, young adult women who are recommended for vaccination demonstrate much lower vaccination rates and higher rates of infection. In a recent Phase I grant, the investigators developed and demonstrated the usability and feasibility of an innovative, culturally-grounded, technology-based narrative intervention that delivers decision narratives in the form of videos via a health kiosk, an underutilized communication strategy for reaching less involved audiences. This brief, low-cost, easily implementable intervention doubled the uptake of the vaccine in a separate pilot study. The proposed Phase II project will: (1) Complete development of the intervention, (2) Evaluate its effectiveness through a randomized clinical trial, and (3) Prepare the product for the market. To accomplish these aims, the investigators will develop the intervention for implementation in waiting rooms as part of check-in procedures. Development includes programming and installing tablets to accomplish these tasks (Aim 1). The investigators will then conduct the evaluation study in four Planned Parenthood clinics in southeastern Pennsylvania (Aim 2). Eligible women will be consented, complete a pretest, and then randomized to view the brief intervention or attention control messages via the tablet. After viewing the messages, the participants will complete a short posttest. Treatment participants will receive follow up texts/emails as reminders to vaccinate, and all participants will receive texts/emails with links that allow completion of posttest surveys at 3- and 9 months. Finally, the investigators will prepare the intervention for the market that includes not only Planned Parenthood but other clinics that are currently served by the project partners as well as the broader market for HPV vaccination (Aim 3). In summary, the proposed communication strategy has wide reaching implications not only for reducing cancer risk, but more broadly for designing brief and easily implemented prevention messages across many domains of public health. The research will also close the health disparities gap in minority, under-served young adult women's access to preventive health care.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking women clients of 4 Planned Parenthood clinics who are between 18 and 26 and have not been vaccinated.

Exclusion Criteria:

* Men, women who do not speak English or are not between 18 and 26 years old, anyone not a client of the 4 Planned Parenthood clinics.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women are the targets for this intervention.
Enrollment: 360 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
HPV Vaccination | 9 months
  Uptake of HPV Vaccine as measured by medical records review and self report

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hecht, Ph.D., Principal Investigator — Real Prevention, LLC
Locations (7):
- United States (7):
  - University of California, Irvine, Irvine, California
  - Planned Parenthood of Illinois, Chicago, Illinois
  - Planned Parenthood of the St. Louis Region and Southwest Missouri, St Louis, Missouri
  - REAL Prevention LLC, Clifton, New Jersey
  - Public Health Management Corporation, Philadelphia, Pennsylvania
  - Planned Parenthood of Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - St. Andrew Development, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Confidential data cannot be shared.

REFERENCES:
- [Background] Hopfer S, Ray AE, Hecht ML, Miller-Day M, Belue R, Zimet G, Evans WD, McKee FX. Taking an HPV vaccine research-tested intervention to scale in a clinical setting. Transl Behav Med. 2018 Sep 8;8(5):745-752. doi: 10.1093/tbm/ibx066. PMID 29425333